CLINICAL TRIAL: NCT01829243
Title: Milnacipran and Neurocognition, Pain and Fatigue in Fibromyalgia: A 13-week Randomized, Placebo Controlled Cross Over Trial
Brief Title: Milnacipran and Neurocognition, Pain and Fatigue in Fibromyalgia : A 13-week Randomized, Placebo Controlled Cross Over Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00026392
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2014-08

CONDITIONS: Fibromyalgia; Neurocognition
Keywords: Milnacipran; Fibromyalgia; Neurocognition
MeSH Terms: conditions — Fibromyalgia | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Milnacipran (Experimental): Eligible subjects will receive milnacipran (12.5 mg-200 mg/day) in the forces titration schedule in flexible doses to the maximum tolerated dose starting with 12.5 mg qd for 1 day, 12.5 mg bid for 2 days, 25 mg bid for 4 days, 50 mg bid for 7 days and 100 mg bid thereafter. Patients who cannot tolerate higher doses will have a step-wise reduction in doses (e.g. 200 mg/day dose will be reduced to 100 mg/day; 100 mg/day will be reduced to 50 mg/day). Drug will be discontinued at the end of the study.
  Interventions: Drug: Milnacipran; Drug: Placebo
- Placebo (Placebo Comparator): Eligible subjects will receive placebo (12.5 mg-200 mg/day) in the forces titration schedule in flexible doses to the maximum tolerated dose starting with 12.5 mg qd for 1 day, 12.5 mg bid for 2 days, 25 mg bid for 4 days, 50 mg bid for 7 days and 100 mg bid thereafter. Patients who cannot tolerate higher doses will have a step-wise reduction in doses (e.g. 200 mg/day dose will be reduced to 100 mg/day; 100 mg/day will be reduced to 50 mg/day). Drug will be discontinued at the end of the study.
  Interventions: Drug: Milnacipran; Drug: Placebo

INTERVENTIONS:
Drug: Milnacipran
  Other Names: Savella
Drug: Placebo

SUMMARY:
This study was designed to investigate whether milnacipran is safe and effective in improving cognitive function in fibromyalgia. In addition, this study was aimed to investigate whether improvement in neurocognitive status due to milnacipran correlates with improvements in pain, to investigate whether improvement in neurocognitive status due to milnacipran correlates with improvements in fatigue, and to determine whether treatment with improvement in neurocognitive status, pain and fatigue correlates with functional improvement.

DETAILED DESCRIPTION:
Cognitive dysfunction is observed in fibromyalgia, especially for episodic memory, learning, and working memory.There is evidence for dysregulation of the attention system from low-level sensory processes up to emotional processes, and increased sensitivity to distraction.Milnacipran's balance of norepinephrine (NE) to serotonin (5-HT) of 3:1, similar to amitriptyline, a tricyclic that has demonstrated efficacy in fibromyalgia, as compared to venlafaxine which is 1:30, or duloxetine which is 1:10.7 In addition, because of milnacipran's effect on 5-HT, it should also be effective in treating other symptoms such as sleep disturbances and mood changes, which are associated to fibromyalgia, as well as other functional somatic syndromes. It is worth noting that several medications to treat fibromyalgia are sedating (e.g pregabalin, opioids, muscle relaxants) and impair neurocognition.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years.
* Specific diagnosis of FM by the participant's rheumatologist or physician, including written confirmation, from a physician, of the FM diagnosis.
* Confirmation of the FM diagnosis by American College of Rheumatology Criteria and a physical tender point examination.
* Ability to give informed consent.
* If female, nonpregnant/nonlactating.
* If a sexually active female of reproductive potential, must be using adequate contraception (i.e., oral contraceptives, barrier protection, or prior tubal ligation) during the trial.

Exclusion Criteria:

* Bipolar disorders, any psychotic disorder.
* the existence of concomitant rheumatological disorders, including rheumatoid arthritis, systemic lupus erythematosus, Hashimoto's disease, Sjogren's syndrome or scleroderma.
* Substance dependence (except nicotine dependence) in the previous 3 months.
* Currently suicidal or high suicide risk.
* Serious or unstable medical disorders.
* Any psychotropic drug treatment in the previous 2 weeks before screening.
* A positive urine pregnancy test.
* Screening laboratory values three times the limits of normal or judged clinically significant by the investigator.
* History of hypersensitivity to milnacipran.
* Seizure disorder, traumatic brain injury, any CNS disorder that affects cognitive status.
* Concomitant meds: A minimum of 30 days on stable dose of analgesics and a minimum of 4 week washout from antidepressants and fibromyalgia specific medication ( e.g. pregabalin, neurontin) and supplements ( St John's wort, SAM-E).
* Narrow angle glaucoma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin A Patkar, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center / Civitan Building, Durham, North Carolina, United States

REFERENCES:
- [Derived] Kim JL, Rele S, Marks DM, Masand PS, Yerramsetty P, Millet RA, Keefe RS, Patkar AA. Effects of milnacipran on neurocognition, pain, and fatigue in fibromyalgia: a 13-week, randomized, placebo-controlled, crossover trial. Prim Care Companion CNS Disord. 2013;15(6):PCC.13m01555. doi: 10.4088/PCC.13m01555. Epub 2014 Dec 26. PMID 24800123

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized to receiving milnacipran-washout-placebo or placebo- washout-milnacipran for 6 weeks, followed by a 1 week washout and then cross over to the other arm for another 6 weeks. The overall trial lasted 13 weeks starting on July 2011 and ending in May 2013.
Groups:
- Milnacipran First, Then Placebo: Patients randomized to receiving milnacipran first.
- Placebo First, Then Milnacipran: Patients randomized to receive placebo first
Period: First Intervention
Arm/Group | Milnacipran First, Then Placebo | Placebo First, Then Milnacipran
Started | 11 | 15
Completed | 7 | 13
Not Completed | 4 | 2
Not completed — Screen Failure | 4 | 2
Period: Washout Period of 1 Week
Arm/Group | Milnacipran First, Then Placebo | Placebo First, Then Milnacipran
Started | 7 | 13
Completed | 7 | 13
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Milnacipran First, Then Placebo | Placebo First, Then Milnacipran
Started | 7 | 13
Completed | 7 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline information is presented for subjects who completed the study.
Arm/Group | Subjects Who Completed the Study
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (9.1)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale for Pain
Description: Visual Analogue Scale for Pain operationally is a 100 mm line anchored by word descriptors at each end. The patient marks a point on the line that reflects their current pain state. The distance in mm from the left anchor point is the score. Higher scores indicate more pain.
Time Frame: Baseline, Week 1, 2,4, and 6 weeks
Population: Analysis employed Intent-to-Treat with Last Observation Carried Forward (LOCF) analysis. The Intent-to-Treat group (ITT) was comprised of all subjects who received at least one dose of the medication.
Measure: Mean (Full Range); unit: mm
Groups:
- Milnacipran: Data is summarize for all patients while they were taking Milnacipran.
- Placebo: Data is summarize for all patients while they were taking the placebo.
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 20 | 20
mm
  Week 0 | 59.4 [4.5 to 59.5] | 68.6 [3.9 to 69.4]
  Week 1 | 58.5 [3.4 to 59.1] | 66.2 [3.4 to 67.3]
  Week 2 | 55.7 [3.0 to 56.3] | 61.5 [3.1 to 62.6]
  Week 4 | 56.9 [2.7 to 57.1] | 54.4 [2.8 to 55.2]
  week 6 | 54.4 [2.7 to 55.9] | 60.4 [2.5 to 60.5]

2. Primary Outcome: Changes in The Fatigue Severity Scale (FSS)
Description: The Fatigue Severity Scale (FSS) is composed of nine items with a seven-point response format. The minimum score = 9 and maximum score possible = 63. Higher scores = greater fatigue severity.
  Sample questions include "I am easily fatigued" and "Exercise brings on my fatigue." In the initial validation study, internal consistency for the Fatigue Severity Scale was high for specific illness groups (MS and lupus) and healthy controls. The scale clearly distinguished patients from controls and it was moderately correlated with a single-item visual analogue scale of fatigue intensity. In all patients, clinical improvement in fatigue was associated with reductions in scores on the Fatigue Severity Scale. The Fatigue Severity Scale is also a practical measure due to its brevity and ease of administration and scoring.
Time Frame: Baseline, Week 1, 2,4, and 6 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale
  Week 0 | 56.3 [44.0 to 56.7] | 49.2 [44.0 to 49.2]
  Week 1 | 54.0 [44.0 to 54.5] | 53.4 [44.0 to 53.6]
  Week 2 | 53.7 [44.0 to 53.7] | 52.2 [44.0 to 52.5]
  Week 4 | 54.1 [44.0 to 54.5] | 52.8 [44.0 to 53.1]
  Week 6 | 52.1 [44.0 to 52.5] | 53.0 [44.0 to 53.7]

3. Primary Outcome: Composite Brief Assessment of Cognition (BAC) Score
Description: The composite BAC score is calculated by scoring each of the 6 individual tests (Verbal Memory Recall, Digit Sequencing, Token Motor Task, Verbal Fluency, Symbol Coding, and Tower of London), comparing each score to a healthy control sample to create z-scores, summing the z-scores, and rescaling the sum. The composite score range is -2127.8 to 1878.8, with higher scores indicating better cognition.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 41.2 (7.3) | 40.9 (10.4)
  Week 6 | 42.9 (8.0) | 42.9 (7.8)

4. Secondary Outcome: MATRICS Consensus Cognitive Battery Composite Score
Description: (MATRICS) Consensus Cognitive Battery measures cognitive functioning within 7 domains: speed of processing, attention/vigilance, working memory (non verbal and verbal), verbal learning, visual learning, reasoning and problem solving and social cognition.
  The composite score is calculated by the MATRICS computer program, which equally weights each of the 7 domain scores. The range of composite scores is 20-80. Higher scores indicate higher levels or cognitive functioning, while lower scores indicate lower levels of cognitive functioning.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Milnacipran: Data is summarize for all patients while they were taking the Milnacipran.
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 41.4 (7.4) | 37.8 (9.6)
  Week 1 | 41.0 (9.7) | 40.6 (10.0)

ADVERSE EVENTS:
Groups:
- Milnacipran: Adverse events in this group occurred while subjects were taking Milnacipran.
- Placebo: Adverse events in this group occurred while subjects were taking Placebo.
Arm/Group | Milnacipran | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 12/20 | 18/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Milnacipran (N=20) | Placebo (N=20)
Depression (Psychiatric disorders) | 2 | 2
Insomnia (General disorders) | 2 | 6
Tiredness (General disorders) | 0 | 1
Pain (General disorders) | 1 | 4
Dizziness (Nervous system disorders) | 1 | 2
Restlessness (Nervous system disorders) | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Appetite change (Metabolism and nutrition disorders) | 1 | 1
Urinary difficulty (Renal and urinary disorders) | 1 | 0
Itching (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes